CLINICAL TRIAL: NCT04343768
Title: An Investigation Into Beneficial Effects of Interferon Beta 1a, Compared to Interferon Beta 1b And The Base Therapeutic Regiment in Moderate to Severe COVID-19: A Randomized Clinical Trial
Acronym: COVIFERON
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Shahid Beheshti University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Seyed Sina Naghibi Irvani, MD, MPH, MBA, Senior Researcher., Dr., Shahid Beheshti University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Different Interferons in COVID
Record Dates: First submitted 2020-04-08; First posted 2020-04-13 (Actual); Last update posted 2020-05-05 (Actual); Status verified 2020-05

CONDITIONS: COVID-19
Keywords: COVID-19; Novel Coronavirus; Interferon Beta 1a; Interferon Beta 1b
MeSH Terms: conditions — COVID-19 | interventions — Hydroxychloroquine; Lopinavir; Interferon beta-1a; Interferon beta-1b

STUDY DESIGN:
Intervention Model Description: The present study is a randomized clinical trial, with the approval of the ethics committee will be conducted on patients who have a positive test confirming COVID-19 in Loghman Hakim Medical Education Center in Tehran. Patients will be randomly assigned to the three arms of the study.
  Patients will be allocated to three therapeutic arms (Hydroxychloroquine + Lopinavir / Ritonavir + Interferon-β 1a group and Hydroxychloroquine + Lopinavir / Ritonavir + Interferon-β 1b group and the Base Therapeutic Regiment Group, i.e., Hydropinchloroquine + / Ritonavir. For this purpose, we will use the method of Balance Block Randomization for three groups.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Hydroxychloroquine + Lopinavir / Ritonavir + Interferon-β 1a (Experimental)
  Interventions: Drug: Hydroxychloroquine; Drug: Lopinavir / Ritonavir; Drug: Interferon Beta-1A
- Hydroxychloroquine + Lopinavir / Ritonavir + Interferon-β 1b (Experimental)
  Interventions: Drug: Hydroxychloroquine; Drug: Lopinavir / Ritonavir; Drug: Interferon Beta-1B
- Control group: hydroxychloroquine + Lopinavir / Ritonavir (Active Comparator)
  Interventions: Drug: Hydroxychloroquine; Drug: Lopinavir / Ritonavir

INTERVENTIONS:
Drug: Hydroxychloroquine — This Drug will be used in all arms.
Drug: Lopinavir / Ritonavir — This Drug will be used in all arms.
Drug: Interferon Beta-1A — This drug will be only used in Arm 1.
  Arms: Hydroxychloroquine + Lopinavir / Ritonavir + Interferon-β 1a
Drug: Interferon Beta-1B — This drug will be only used in Arm 2.
  Arms: Hydroxychloroquine + Lopinavir / Ritonavir + Interferon-β 1b

SUMMARY:
The present study is a randomized clinical trial, with the approval of the ethics committee will be conducted on patients who have a positive test confirming COVID-19 in Loghman Hakim Medical Education Center in Tehran. Patients will be randomly assigned to the three arms of the study and after completing the course of treatment and collecting and analyzing the necessary information from each patient, the results of the study will be published both on this site and in the form of an article in a reputable international journal.

DETAILED DESCRIPTION:
According to previous studies, IFN-β has strong antiviral activity and also has an acceptable safety profile. Based on possible therapeutic effects, We decided to lead An Investigation into Beneficial Effects of Interferon Beta 1a, Compared to Interferon Beta 1b And The Base Therapeutic Regiment in Moderate to Severe COVID-19. In a 2003 study, SARS was treated with different human interferons and found that IFN-β was 5 to 10 times more effective than other types of interferons and the strongest antiviral drug possible against SARS-CoV.

The present study is a randomized clinical trial, with the approval of the ethics committee will be conducted on patients who have a positive test confirming COVID-19 in Loghman Hakim Medical Education Center in Tehran.

Patients will be allocated to three therapeutic arms (Hydroxychloroquine + Lopinavir / Ritonavir + Interferon-β 1a group and Hydroxychloroquine + Lopinavir / Ritonavir + Interferon-β 1b group and the Base Therapeutic Regiment Group, i.e., Hydropinchloroquine + / Ritonavir. For this purpose, we will use the method of Balance Block Randomization for three groups.

After completing the course of treatment and collecting and analyzing the necessary information from each patient, the results of the study will be published both on this site and in the form of an article in a reputable international journal.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18
* COVID-19 Confirmed Cases By Means of RT-PCR
* Oxygen saturation (SPO2) ≤ 93% OR respiratory rate ≥ 24
* At least one of the following: Calibrated contactless infrared forehead thermometry temperature of ≥37.8, cough, sputum production, nasal discharge, myalgia, headache or fatigue on admission.
* Time of onset of the symptoms should be acute ( Days ≤ 14)

Exclusion Criteria:

* Refusal to participate expressed by patient or legally authorized representative if they are present
* Patients with prolonged QT or PR intervals, Second or Third Degree heart block, Arrhythmias including torsade de pointes
* Patients using drugs with potential interaction with Hydroxychloroquine + Lopinavir/Ritonavir, Interferon-β 1a، Interferon-β 1b.
* Pregnant or lactating women.
* History of alcohol or drug addiction in the past 5 years.
* Blood ALT/AST levels > 5 times the upper limit of normal on laboratory results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2020-04-09 (Actual); Primary Completion 2020-04-27 (Actual); Study Completion 2020-04-27 (Actual)

PRIMARY OUTCOMES:
Time to clinical improvement | From date of randomization until 14 days later.
  Improvement of two points on a seven-category ordinal scale (recommended by the World Health Organization: Coronavirus disease (COVID-2019) R&D. Geneva: World Health Organization) or discharge from the hospital, whichever came first.

SECONDARY OUTCOMES:
Mortality | From date of randomization until 14 days later.
  If the patient dies, we have reached an outcome.
SpO2 Improvement | Days 1, 2, 3, 4, 5, 6, 7 and 14.
  Pulse-oxymetry
Incidence of new mechanical ventilation use | From date of randomization until 14 days later.
  Incidence of new mechanical ventilation use
Duration of hospitalization | From date of randomization until the date of hospital discharge or date of death from any cause, whichever came first, assessed up to 14 days.
  Duration of hospitalization (days)

CONTACTS AND LOCATIONS:
Overall Officials: Ilad Alavi Darazam, MD, Study Chair — Shahid Beheshti University of Medical Sciences; Shervin Shokouhi, MD, Study Director — Shahid Beheshti University of Medical Sciences; Minoosh Shabani, MD, Principal Investigator — Shahid Beheshti University of Medical Sciences; Mohammadreza Haji Esmaelie, MD, Principal Investigator — Shahid Beheshti University of Medical Sciences; Seyed Sina Naghibi Irvani, MD, MPH, MBA, Principal Investigator — Shahid Beheshti University of Medical Sciences
Locations (1):
- Loghman Hakim Hospital, Shahid Beheshti University of Medical Sciences and Health Services, Tehran, Iran

IPD SHARING:
Plan to Share IPD: Yes
One year after the publication of the results in a journal, Qualifying researchers who reach out to Dr. Seyed Sina Naghibi Irvani at "sina.irvani@sbmu.ac.ir" or "sina.irvani@gmail.com" and submit a proposal with a valuable research question can have access to data and supporting information.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: One year after the publication of the results in a journal.
Access Criteria: Qualifying researchers who reach out to Dr. Seyed Sina Naghibi Irvani at "sina.irvani@sbmu.ac.ir" or "sina.irvani@gmail.com" and submit a proposal with a valuable research question.

REFERENCES:
- [Background] Zu ZY, Jiang MD, Xu PP, Chen W, Ni QQ, Lu GM, Zhang LJ. Coronavirus Disease 2019 (COVID-19): A Perspective from China. Radiology. 2020 Aug;296(2):E15-E25. doi: 10.1148/radiol.2020200490. Epub 2020 Feb 21. PMID 32083985
- [Background] Lu R, Zhao X, Li J, Niu P, Yang B, Wu H, Wang W, Song H, Huang B, Zhu N, Bi Y, Ma X, Zhan F, Wang L, Hu T, Zhou H, Hu Z, Zhou W, Zhao L, Chen J, Meng Y, Wang J, Lin Y, Yuan J, Xie Z, Ma J, Liu WJ, Wang D, Xu W, Holmes EC, Gao GF, Wu G, Chen W, Shi W, Tan W. Genomic characterisation and epidemiology of 2019 novel coronavirus: implications for virus origins and receptor binding. Lancet. 2020 Feb 22;395(10224):565-574. doi: 10.1016/S0140-6736(20)30251-8. Epub 2020 Jan 30. PMID 32007145
- [Background] Chen Y, Liu Q, Guo D. Emerging coronaviruses: Genome structure, replication, and pathogenesis. J Med Virol. 2020 Apr;92(4):418-423. doi: 10.1002/jmv.25681. Epub 2020 Feb 7. PMID 31967327
- [Background] Spiegel M, Pichlmair A, Muhlberger E, Haller O, Weber F. The antiviral effect of interferon-beta against SARS-coronavirus is not mediated by MxA protein. J Clin Virol. 2004 Jul;30(3):211-3. doi: 10.1016/j.jcv.2003.11.013. PMID 15135736
- [Background] Channappanavar R, Perlman S. Pathogenic human coronavirus infections: causes and consequences of cytokine storm and immunopathology. Semin Immunopathol. 2017 Jul;39(5):529-539. doi: 10.1007/s00281-017-0629-x. Epub 2017 May 2. PMID 28466096
- [Background] Cinatl J, Morgenstern B, Bauer G, Chandra P, Rabenau H, Doerr HW. Treatment of SARS with human interferons. Lancet. 2003 Jul 26;362(9380):293-4. doi: 10.1016/s0140-6736(03)13973-6. PMID 12892961
- [Background] Hensley LE, Fritz LE, Jahrling PB, Karp CL, Huggins JW, Geisbert TW. Interferon-beta 1a and SARS coronavirus replication. Emerg Infect Dis. 2004 Feb;10(2):317-9. doi: 10.3201/eid1002.030482. PMID 15030704
- [Background] Zeng YM, Xu XL, He XQ, Tang SQ, Li Y, Huang YQ, Harypursat V, Chen YK. Comparative effectiveness and safety of ribavirin plus interferon-alpha, lopinavir/ritonavir plus interferon-alpha, and ribavirin plus lopinavir/ritonavir plus interferon-alpha in patients with mild to moderate novel coronavirus disease 2019: study protocol. Chin Med J (Engl). 2020 May 5;133(9):1132-1134. doi: 10.1097/CM9.0000000000000790. No abstract available. PMID 32149772
- [Derived] Alavi Darazam I, Shokouhi S, Pourhoseingholi MA, Naghibi Irvani SS, Mokhtari M, Shabani M, Amirdosara M, Torabinavid P, Golmohammadi M, Hashemi S, Azimi A, Jafarazadeh Maivan MH, Rezaei O, Zali A, Hajiesmaeili M, Shabanpour Dehbsneh H, Hoseyni Kusha A, Taleb Shoushtari M, Khalili N, Soleymaninia A, Gachkar L, Khoshkar A. Role of interferon therapy in severe COVID-19: the COVIFERON randomized controlled trial. Sci Rep. 2021 Apr 13;11(1):8059. doi: 10.1038/s41598-021-86859-y. PMID 33850184
- [Derived] Irvani SSN, Golmohammadi M, Pourhoseingholi MA, Shokouhi S, Darazam IA. Effectiveness of Interferon Beta 1a, compared to Interferon Beta 1b and the usual therapeutic regimen to treat adults with moderate to severe COVID-19: structured summary of a study protocol for a randomized controlled trial. Trials. 2020 Jun 3;21(1):473. doi: 10.1186/s13063-020-04382-3. PMID 32493468
- See also: Related Info — https://doi.org/10.1101/2020.02.03.20020263